CLINICAL TRIAL: NCT02686112
Title: Pregnancy Outcome in Woman With Threatened Abortion
Acronym: POTA
Status: Completed | Type: Observational
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, Eyal.levy, Dr., Bnai Zion Medical Center
Other Study IDs: BNZ-0043-14
Record Dates: First submitted 2016-01-28; First posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Threatened Abortion
MeSH Terms: conditions — Abortion, Threatened

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study aims to quantify the relations between first & second trimester bleeding and maternal & neonatal morbidity. Additionally, the study will help in assessing the risk for abortions in women with threatened abortions and the risk factors for threatened abortion.

DETAILED DESCRIPTION:
the study is following woman retrospectively through their pregnancy from the first trimester troughout delivery .

we will measure the relation between first and/or second trimester bleeding ( threatend abortion ) and pregnancy outcome ( as written below ) - maternal and neonatal .

ELIGIBILITY:
Inclusion Criteria:

* Women who attended the Emergency department with vaginal bleeding and/or abdominal pain and were on their 20th week of pregnancy or less.

Exclusion Criteria:

* Women with any background that can explain vaginal bleeding or any other circumstance that can explain it.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women who attanded the Emergency department with vaginal bleeding and/or abdominal pain and were on their 20th week of pregnancy or less.
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2007-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Maternal and neonatal outcome in pregnancies with 1st and 2nd trimester bleeding | 9 months
  by using our data in the past 7 years we will examine retrospectively cases of patients from their first admission due to vaginal bleeding throgh their pregnancy and labor .
  the mesearment will include : Intra uterine growth retardation , Antepartum hemorrhage, premature rupture of membrane, Intra uterine fetal death , Preterm delivery, Apgar less than 7, Congenital malformation, Mode of delivery - vaginal delivery vs. cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Levy, Resident, Principal Investigator — Bnai Zion

IPD SHARING:
Plan to Share IPD: No